CLINICAL TRIAL: NCT03407001
Title: Lesion Detection in Cirrhotic Patients With Contrast Enhanced Ultrasound and the Accuracy of Contrast Enhanced Ultrasound Li-RADS for Hepatocellular Carcinoma Diagnosis
Brief Title: Contrast Enhanced Ultrasound With Lumason in Detecting Liver Cancer in Participants With Cirrhosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017-0691; NCI-2018-00895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0691 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); R01CA195524 (NIH)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Screening (US, CEUS, Lumason) (Experimental): Within 30 days of routine MRI, participants undergo non-contrast ultrasound of the abdomen. Participants then receive Lumason IV and undergo contrast-enhanced ultrasound of the abdomen over 1 hour in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Contrast-Enhanced Ultrasound; Drug: Sulfur Hexafluoride Lipid Microspheres; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Contrast-Enhanced Ultrasound — Undergo CEUS
  Other Names: CEUS
Drug: Sulfur Hexafluoride Lipid Microspheres — Given IV
  Other Names: Lumason; SF6 Lipid Microspheres; Sulfur Hexafluoride Lipid-type A Microspheres
Procedure: Ultrasound — Undergo non-contrast US

SUMMARY:
This early phase I trial studies how well contrast enhanced ultrasound with sulfur hexafluoride lipid microspheres (Lumason) works in detecting liver cancer in participants with cirrhosis. Contrast enhanced-ultrasounds use contrast agents, such as Lumason, that are injected into a vein in order to help certain organs and tissues show up more clearly on scans. Contrast enhanced ultrasound with Lumason may help doctors more easily find liver cancer compared to ultrasounds without contrast agent.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the accuracy of contrast enhanced ultrasound (CEUS) utilizing contrast agent sulfur hexafluoride lipid-type A microspheres compared to B-mode non-contrast enhanced ultrasound for liver lesion detection, including hepatocellular carcinoma (HCC), in cirrhotic ultrasound (US) patients.

SECONDARY OBJECTIVES:

I. Determine the concordance of CEUS vs. contrast enhanced magnetic resonance imaging (CE-MRI) Liver Imaging Reporting and Data Systems (Li-Rads).

OUTLINE:

Within 30 days of routine MRI, participants undergo non-contrast ultrasound of the abdomen. Participants then receive Lumason intravenously (IV) and undergo contrast-enhanced ultrasound of the abdomen over 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Diagnosis of cirrhosis based on one or more of the following: histology, US, computed tomography (CT) or MRI showing cirrhosis, +/- lesions seen on CE-MRI

Exclusion Criteria:

* History of hypersensitivity to sulfur hexafluoride lipid microsphere components or to any of the inactive ingredients in Lumason
* Pregnant patients-excluded by history
* Pediatric patients, as pediatric cirrhosis is uncommon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of contrast enhanced ultrasound (CEUS) with contrast agent sulfur hexafluoride lipid-type A microspheres and B-mode non-contrast enhanced ultrasound | Up to 3 years
  The study will estimate the sensitivity of ultrasound (US) and CEUS in patients with detectable lesions on magnetic resonance imaging (MRI). The analysis will be conducted at the patient level with a binary outcome of 0 if the patient has no detectable lesions and 1 if the patient has one or more detectable lesions. The study will use McNemar's test to compare US vs. CEUS in patients with any detectable lesions on MRI. The test assesses whether the two tests have equivalent marginal probabilities (i.e. probability of detecting at least one lesion with US and CEUS is equivalent). McNemar's test statistic depends only on patients where US and CEUS disagree.

SECONDARY OUTCOMES:
Assessment of CEUS and contrast enhanced magnetic resonance imaging (CE-MRI) Liver Imaging Reporting and Data Systems (Li-Rads) | Up to 3 years
  The study will assess the concordance between CEUS Li-Rads and MRI Li-Rads scoring results for each lesion using a multinomial logit random effects model. The study will summarize the characteristics (the size, location, vascularity and enhancement pattern) of lesions detected by only one imaging modality, stratified by imaging type.

CONTACTS AND LOCATIONS:
Overall Officials: Ott Le, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org